CLINICAL TRIAL: NCT00006493
Title: Rosiglitazone in the Treatment of HIV-Associated Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00096-1006; M01RR000096 (NIH)
Record Dates: First submitted 2000-11-14; First posted 2000-11-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: HIV Infections; Hyperlipidemia
Keywords: HIV-associated hyperlipidemia
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The purpose of this research is to study the effects of rosiglitazone, a drug usually taken for Type II diabetes, on HIV-associated hyperlipidemia. HIV-associated lipodystrophy is a medical condition characterized by gradual changes in the distribution of body fat. The body fat located in the extremities and face disappears while body fat around the abdomen and upper back increases. Certain biochemical changes occur in association with these changes in fat distribution. Lipid levels particularly serum triglycerides are increased. HDL, the "good cholesterol" is decreased. Higher than normal level of insulin or insulin resistance is also found in this condition. This latter condition is one of the hallmarks of Type II diabetes. The protease inhibitors, a class of HIV medications, are associated with the occurrence of HIV-associated lipodystrophy. It has been suggested that a biochemical pathway known as the peripheral peroxisomal activating receptor (PPAR) gamma system is blocked leading to the onset of this condition.

Rosiglitazone is a new drug approved by the FDA in 1999 for the treatment of type II diabetes. It lowers blood sugar by improving insulin resistance, which as mentioned before, is the hallmark of Type II diabetes. It has also been noted to improve blood lipid levels. Rosiglitazone works by stimulating the PPAR gamma system. It is hoped that this drug can turn on the PPAR system and reverse the HIV-associated lipodystrophy syndrome.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive with CD4 count > 500 and undetectable viral load
* Treated with protease inhibitors for more than three months
* Serum triglycerides > 400mg/dl
* Clinical diagnosis of HIV-associated lipodystrophy
* No history of type II diabetes
* Fasting blood sugar < 126 mg/dl
* No history of liver disease
* Negative Hepatitis B antigen and Hepatitis C antibody
* Not on the following medications: warfarin, digoxin, nifedipine, erythromycin, cyclosporine or HMG coA-reductase inhibitors
* Hemoglobin > 11g/dl
* Women of childbearing age must consent to barrier contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, New York, New York, United States